CLINICAL TRIAL: NCT01090609
Title: Multicenter, Prospective, Non-randomized Study to Evaluate the Safety of Cronus® Cobalt Chromium Coronary Stent - Study After 9 Months
Brief Title: Study to Evaluate the Safety of Cronus® - Cobalt Chromium Coronary Stent
Acronym: CRONUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scitech Produtos Medicos Ltda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Scitech 002
Record Dates: First submitted 2010-03-18; First posted 2010-03-22 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Stent; Cobalt-Chromium coronary stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stent implantation (Experimental): Cronus Stent implantation
  Interventions: Device: Stent implantation

INTERVENTIONS:
Device: Stent implantation — Stent implantation
  Other Names: Angioplasty

SUMMARY:
The objective this study is evaluate the performance and safety of Chronus® cobalt-chromium coronary stent in patients with "de novo" native coronary artery lesions treated with 19-mm-long stents in long-term 9 months.

DETAILED DESCRIPTION:
The use of coronary stents has optimized the results of coronary balloon angioplasty for two reasons:

1. reduced acute complications, such as acute and subacute occlusion, as well as the need of urgent myocardial revascularization;
2. reduced coronary restenosis. STRESS and BENESTENT 1 pivotal clinical trials7,9 laid the foundations for approval and confirmation of the efficacy of coronary stents. These studies showed a reduction in the binary angiographic restenosis rates from 42.1% to 31.6% (p<0.05) and from 32% to 22% (p=0.02), respectively. The efficacy of coronary stents is due to the fact that these devices reduce the acute elastic recoil and late negative remodeling of coronary arteries because of their capacity to maintain the vessel adequately open without reducing vessel diameter.

Cronus® stent is fabricated in cobalt-chromium. This alloy is currently used cardiovascular stents and permanent implants in orthopedic (hips, knees), dental and maxillofacial surgeries. Guidant and Medtronic have conducted clinical evaluations of stents fabricated with a similar cobalt-chromium alloy and demonstrated safety and efficacy of the investigational devices. Both stents are currently available in the European market.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤75 years;
2. Symptomatic cardiac ischemic disease and/or documented evidence of myocardial ischemia;
3. Types B1 and B2 coronary lesions (according to the ACC/AHA classification modified by Ellis);
4. Target lesion located in a native coronary artery;
5. Target lesion in vessel with diameter ranging from 2.5 to 3.5 mm (by visual estimate) amenable to treatment (coverage) with a 19-mm-long stent;
6. Target lesion with >50% diameter stenosis (by visual estimate);
7. Acceptable candidate to myocardial revascularization surgery (coronary artery bypass graft surgery);
8. The subject has been fully informed of the nature of the study, is willing to comply with all study requirements and will provide written informed consent as approved by the Ethics Committee of the respective clinical site.

Exclusion Criteria:

1. Female patients of childbearing potential;
2. Recent Q-wave myocardial infarction occurred within 48 hours prior to the index procedure. Recent Q-wave or non-Q-wave myocardial infarction with still elevated levels of cardiac markers;
3. Documented left ventricular ejection fraction <30%;
4. Renal dysfunction (creatinine > 2.0 mg/dL or 177 µmol/L);
5. Platelet count <100,000 cells/mm³ or >700,000 cells/mm³.;
6. White blood cell count <3,000 cells/mm3;
7. Suspected or documented hepatic disease (including laboratorial evidence of hepatitis);
8. Heart transplant receptor;
9. Known hypersensitivity to cobalt-chromium or to medications such as aspirin, clopidogrel bisulfate (Plavix or ISCOVER), ticlopidine (Ticlid) or heparin.
10. Concurrent medical condition with a life expectancy of less than 12 months;
11. Any major medical condition that, in the Investigator's opinion, may interfere with the optimal participation of the patient in this study;
12. Subject is currently participating in an investigational drug or another device study, including planned participation in an investigational drug or another device study during the course of the present investigation;
13. Coronary angioplasty (with or without stenting) less than 9 months before the index procedure at any site of the target vessel;
14. Previous coronary angioplasty (with or without stenting) at any time (>9 months) in a vessel segment less than 5 mm proximal or distal to the target lesion.
15. Planned coronary angioplasty (with or without stenting) in the first 12 months after the index procedure in any segment of the target vessel;

Angiography Exclusion Criteria:

1. Restenotic target lesion;
2. More than one lesion requiring treatment in the same vessel;
3. Target vessel diameter <2.5 mm or >3.5 mm (by visual estimation);
4. Long target lesion not amenable to treatment (coverage) with a 19-mm-long stent;
5. Unprotected coronary artery branch lesion (≥50% diameter stenosis)
6. Target lesion is located in a surgical bypass graft;
7. Total vessel occlusion (TIMI flow grade 0-1);
8. Target lesion with ostial location;
9. Target lesion located in a lateral branch bifurcation >2.5mm or requiring lateral branch stenting;
10. Calcified target lesion that anticipates unsuccessful/impracticable predilation;
11. Target vessel with excessive tortuosity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2010-05; Primary Completion 2012-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Clinical Follow-up | 30 days after the procedure
  All patients are invited to return for a clinical visit at 30 days post-procedure to evaluate possible adverse events and on the continuity of cardiac medication.

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Feres, Medicine, Principal Investigator — Instituto Dante Pazzanese de Cardiologia
Locations (13):
- Brazil (13):
  - Hospital São Salvador Goiânia, Goiânia, Goiás
  - Hospital Santa Genoveva, Goiânia, Goiás
  - Irmandade Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital Santa Isabel, Blumenau, Santa Catarina
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - Instituto de Assistência Médica ao Servidor Público Estadual - Iamspe, São Paulo, São Paulo
  - Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo
  - Hospital São Paulo - UNIFESP, São Paulo, São Paulo
  - São Bernardo Apart Hospital, Colatina - ES
  - Santa Casa de Franca, Franca - SP
  - Hospital Vera Cruz, Patos de Minas - MG
  - Instituto de Medicina Integral Professor Fernando Figueira - IMIP, Recife - PE
  - Santa Casa de Misericórdia de São José do Rio Preto, São José Do Rio Preto - SP

REFERENCES:
- See also: Sponsor site — http://www.scitechmed.com
- See also: National Information System on Ethics in Research involving Human — http://portal2.saude.gov.br/sisnep